CLINICAL TRIAL: NCT06561061
Title: Zinc for Infection Prevention in Sickle Cell Anemia-2
Brief Title: Zinc for Infection Prevention in Sickle Cell Anemia-2 (ZIPS-2)
Acronym: ZIPS-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Global Health Uganda LTD (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Chandy John, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-841
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease
Keywords: Zinc; All-cause infections
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: A randomized double-blinded placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc (Experimental): Dispersible zinc sulfate tablet (20 mg)
  Interventions: Drug: zinc sulfate
- Placebo (Placebo Comparator): Dispersible identical placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zinc sulfate — Dispersible (20 mg) tablet
  Arms: Zinc
Drug: Placebo — Dispersible tablet
  Arms: Placebo

SUMMARY:
A randomized double-blinded placebo-controlled trial of zinc to reduce the incidence of severe or invasive infections in Ugandan children with sickle cell anemia (SCA)

DETAILED DESCRIPTION:
The study will be a randomized, placebo-controlled, double blind clinical trial in which 100 Ugandan children 1.00-4.99 years of age with SCA will receive zinc (20 mg oral dispersible tablet daily) or placebo (identical to zinc in appearance) for 6 months. The primary study outcome will be incidence of infection (all causes).

ELIGIBILITY:
Inclusion Criteria:

* Documented sickle cell anemia (HbSS supported by hemoglobin electrophoresis)
* Age range of 1.00-4.99 years, inclusive, at the time of enrollment
* Weight at least 5.0 kg at the time of enrollment
* Willingness to comply with all study-related treatments, evaluations, and follow-up
* Children whose parents or guardians give full written informed consent

Exclusion Criteria:

* Known other chronic medical condition (e.g., HIV, malignancy, active clinical tuberculosis)
* Severe malnutrition determined by impaired growth parameters as defined by WHO (weight for length/height or height for age z-score <-3, using WHO growth standards)
* Absolute neutropenia (absolute neutrophil count <500)

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of all-cause infections in the zinc vs. placebo groups | 6 months
  Will assess the difference in the incidence of all cause infection between the Placebo arm and the experimental arm

SECONDARY OUTCOMES:
Incidence of infections requiring hospitalization | 6 months
  Incidence of Advance events greater or equal to grade 3
Incidence of adverse events requiring discontinuation of study drug | 6 months
  Incidence of Zinc related Advance events
Incidence of stroke or death | 6 months
  Incidence of death and stroke

OTHER OUTCOMES:
Change in Transcranial Doppler (TCD) velocity from enrollment to 6-month study endpoint | 6 months
  Change in TCD Velocity

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C John, MD, Principal Investigator — Indiana University
Locations (1):
- Jinja Hospital, Jinja, Uganda

IPD SHARING:
Plan to Share IPD: No